CLINICAL TRIAL: NCT01010815
Title: Metagenomic Analysis of Gut Microbiome in Korean Patients With Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Joo Sung Kim, Seoul National University Hospital
Other Study IDs: Gut Microbiome in UC Patients
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; gut microbiome; metagenomics
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will need to give stool samples and colorectal biopsy specimens on 1 or 2 separate occasions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- UC group: clinically and microscopically confirmed UC patients between the age of 19 and 75 years
  Interventions: Procedure: colonoscopy biopsy; Other: stool collection
- Control group: normal healthy controls
  Interventions: Procedure: Colonoscopy biopsy; Other: stool collection

INTERVENTIONS:
Procedure: Colonoscopy biopsy — Colonoscopy biopsy will be performed in rectum, ascending and descending colon at study entry
  Groups: Control group
Other: stool collection — Stool will be collected from participants at study entry
  Groups: Control group
Procedure: colonoscopy biopsy — colonoscopy biopsy will be conducted in rectum, ascending and descending colon from participants 2 times during study - at active phase and inactive phase
  Groups: UC group
Other: stool collection — stool will be collected from participants 2 times during study - at active phase and inactive phase
  Groups: UC group

SUMMARY:
The researchers will investigate gut microbiome in Korean patients with ulcerative colitis and normal control subjects using metagenomic analysis to elucidate the significant difference between two groups This study will help to understand the association between gut microbiome and inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 19 and 75 years
* willing to consent/undergo necessary procedures
* clinically active or inactive Ulcerative colitis

Exclusion Criteria:

* Inability to provide informed consent or
* Clinically severe or fulminant ulcerative colitis
* Previous abdominal surgery
* Pregnancy
* Clinically or laboratory-confirmed gastroenteritis for at least 3 months before sampling
* the use of antibiotics in the past a month before sampling
* the use of probiotics in the past a month before sampling
* Severe cardiovascular or pulmonary disease
* Severe convulsive disorder and current use of anti-convulsive medication
* Malignancy
* Transplantation

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: gastroenterology clinic at SNUH(Seoul National University Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
characterize the difference in gut microbiomes through metagenomic analysis between UC patients and normal control subjects | 1 year

SECONDARY OUTCOMES:
characterize the difference in gut microbiomes through metagenomic analysis between stool specimens and biopsy specimens in participants with UC and normal subjects | 1 year
characterize the difference in gut microbiomes among colonoscopy biopsy locations (rectum, ascending and descending colon) | 1 year
characterize the difference in gut microbiomes between active and inactive UC patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joo Sung Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea